CLINICAL TRIAL: NCT04488484
Title: Medical and Serological Follow-up of the Staff of the Paris Saint-Joseph Hospital Group
Brief Title: Medical and Serological Follow-up of the Staff of the Paris Saint-Joseph Hospital Group Infected With Severe Acute Respiratory Syndrome Coronavirus 2.
Acronym: PERSO-COVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PERSO-COVID
Record Dates: First submitted 2020-07-20; First posted 2020-07-28 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: COVID-19
Keywords: COVID-19; coronavirus; SARS-CoV2
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: The research is a prospective, follow-up cohort, non-randomized and interventional study that aims at following patients who presented a positive serology for the COVID-19
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm (Other): Serology test results
  The Paris Saint- Joseph Hospital Group staff was submitted to a 2 times serology test: the 1st took place between April, 20th to May, 12th and the second, between May, 26th to June, 12th. The employees presenting positive antibodies titers to SARS-CoV-2 will be contacted and asked for a 12 month follow-up study organized by the Occupational Health Team and the team of COVID-19 Serology referents appointed to carry out and coordinate the procedure. Each enrolled member will receive a letter with containing an information letter describing the study with a written consent form and a questionnaire enabling the data to be collected individually on the COVID-19 infection.
  Interventions: Other: Serology test follow-up

INTERVENTIONS:
Other: Serology test follow-up — The enrolled participants will be invited to visit ESS. They will then meet the occupational physician, who wil obtain their free, informed and written consent. The information and consent will be recorded in the personal medical follow-up file.The staff will then complete the self-questionnaire and the ESS physician will provide a prescription for the blood samples to be taken.
  In case of positive answers to one or more of the questions in this self-questionnaire, the enrolled participant will be contacted in order to schedule another post-COVID-19 consultation with additional examinations if needed (new COVID PCR, scanner, etc.).

SUMMARY:
The Coronavirus SARS CoV-2 (COVID-19) pandemic is causing a major global health crisis that is disrupting our hospital organizations and creating potential infectious risks for hospital staff on the front line when it comes to the support of infected people.

In this context, the Paris Saint-Joseph Hospital Group (GhPSJ) very early on wanted to implement an institutional approach aimed, on the one hand, at enabling each of its employees at its two sites (Hôpital Paris Saint-Joseph (HPSJ), Paris 14ème and Hôpital Marie Lannelongue (HML), Le Plessis Robinson, 92) to access their serological status with regard to SARS-CoV-2 and, on the other hand, to identify the risk factors for contracting COVID-19.

This collective approach consisted of an evaluation of its professional practices aimed at assessing the protective measures put in place to protect hospital personnel and identifying sources of potential improvement in the management of the infectious risk required to put in place in case of upcoming COVID-19 cases or any other epidemics in the future.

DETAILED DESCRIPTION:
This institutional process had been validated by senior management and staff representative bodies. It was based on voluntary work, anonymity, the confidential aspect of the employees' analyses with the establishment of a follow-up and an individual counselling organized by the Occupational Health Service (SST) team and a team of COVID-19 Serology referents appointed to carry out and coordinate this process. Among the 3,600 GhPSJ employees, 3,062 (85%) samples were taken (and 404 employees from partner establishments in the hospital complex) for an initial serology test between April, 20th and May,15th and a second test one month later (M1) between May 18th and June 12th. The purpose of this second sampling was to get rid of the fear of another infection that might have occurred on the date of the first serology, and to observe the evolution between the two samples at the end of the epidemic phase.

The first results identified 310 people (231 from the HPSJ site and 56 from the HML site) (10.1%) with a positive serology for SARS CoV-2. However, it was observed that the people infected by the COVID-19, had highly variable IgG antibody titers and these titers changed unexpectedly. In fact, the majority of cases (89%) showed a drop in antibody titers as early as the first month and 20 of them (6.4%) even showed a negativation based on the index of quantitative ELISAs performed.

After only 5 months of hindsight in the face of this new pandemic, there are a few robust and specific data on the immune response following the COVID-19 and its involvement in the clinical impact on infected patients. In addition to the epidemiological interest and potential protection, the use of the immune response is an important therapeutic issue that is currently being evaluated, whether for passive immunization or primary prevention, with highly anticipated prospects for vaccination of populations.

It should be noted that the severely infected patients present characteristics unique to COVID-19 that are rarely seen in other respiratory viral infections, such as severe lymphopenia and eosinopenia, pneumonia and extensive lung damage, cytokine storm leading to acute respiratory distress syndrome and multisystem failure, and numerous atypical presentations (ENT, digestive, mucocutaneous, etc.). A high viral load at the time of first infection and/or repeated exposures to the virus, particularly for healthcare professionals, may be an important factor in the evolution of the disease (severe clinical forms, delayed clinical signs and particular serological kinetics).

In this context, the team in charge of coordinating the institutional project, in connection with the Occupational Health Service (SST) which followed all the personnel exposed during the epidemic period, wishes to propose to the GhPSJ personnel who desires a longitudinal follow-up as part of a research approach aimed at describing the kinetics of the antibodies produced following a COVID-19 infection and a medical follow-up including a self-questionnaire and a consultation specifically targeting the delayed clinical presentations after COVID-19 accompanied by a longitudinal serological follow-up over a longer period.

ELIGIBILITY:
Inclusion Criteria:

* employee aged over 18 years
* employee who participated to the serology tests
* employee who was tested positively to the Covid-19 serology test
* French speaking employee
* employee affiliated to a French social security or any other health insurance system.
* employee who is able to give its free and written consent.

Exclusion Criteria:

* employee under guardianship or curatorship
* employee deprived of liberty
* employee under the protection of justice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-05-23 (Actual)

PRIMARY OUTCOMES:
Immune Response description | 1 month
  The research will describe and distinguish the type of immune response observed both on the basis of the titers of antibodies (IgG and IgM) produced.
Evolution of the SARS-CoV2 overtime | 1 month (after the 1st serology test results)
  the serology test will observe the evolution of the COVID-19 over time, its impact on the staff infected and the memory carried by the associated cellular reaction.

SECONDARY OUTCOMES:
Clinical and Immunological Analysis | 2 months
  the research will focus on the analysis of the hanges in antibody titers over time as a function of the clinical signs observed at initial diagnosis and the post-COVID-19 symptoms and the possible reinfections.
Comparison of the occurrence of clinical events with other immunological data | 2 months
  It will also confront the occurrence of clinical events (post-COVID-19 symptoms and reinfections) with immunological data (antibody levels, cellular immune response) and compare anti-SARS-CoV-2 antibody titers to those determined for other similar viruses (Rubella, Mumps).

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Janice Oh HL, Ken-En Gan S, Bertoletti A, Tan YJ. Understanding the T cell immune response in SARS coronavirus infection. Emerg Microbes Infect. 2012 Sep;1(9):e23. doi: 10.1038/emi.2012.26. Epub 2012 Sep 5. PMID 26038429
- [Background] Li G, Fan Y, Lai Y, Han T, Li Z, Zhou P, Pan P, Wang W, Hu D, Liu X, Zhang Q, Wu J. Coronavirus infections and immune responses. J Med Virol. 2020 Apr;92(4):424-432. doi: 10.1002/jmv.25685. Epub 2020 Feb 7. PMID 31981224
- [Background] Rajendran K, Krishnasamy N, Rangarajan J, Rathinam J, Natarajan M, Ramachandran A. Convalescent plasma transfusion for the treatment of COVID-19: Systematic review. J Med Virol. 2020 Sep;92(9):1475-1483. doi: 10.1002/jmv.25961. Epub 2020 May 12. PMID 32356910
- [Background] Prompetchara E, Ketloy C, Palaga T. Immune responses in COVID-19 and potential vaccines: Lessons learned from SARS and MERS epidemic. Asian Pac J Allergy Immunol. 2020 Mar;38(1):1-9. doi: 10.12932/AP-200220-0772. PMID 32105090
- [Background] Salje H, Tran Kiem C, Lefrancq N, Courtejoie N, Bosetti P, Paireau J, Andronico A, Hoze N, Richet J, Dubost CL, Le Strat Y, Lessler J, Levy-Bruhl D, Fontanet A, Opatowski L, Boelle PY, Cauchemez S. Estimating the burden of SARS-CoV-2 in France. Science. 2020 Jul 10;369(6500):208-211. doi: 10.1126/science.abc3517. Epub 2020 May 13. PMID 32404476
- [Result] Pilmis B, Elkaibi I, Pean de Ponfilly G, Daikha H, Bouzid A, Guihot A, Castreau N, Pradere P, Ketatni H, Mondragon A, Hayem G, Le Pavec J, Laplanche S, Le Monnier A. Evolution of anti-SARS-CoV-2 immune response in a cohort of French healthcare workers followed for 7 months. Infect Dis Now. 2022 Mar;52(2):68-74. doi: 10.1016/j.idnow.2022.01.004. Epub 2022 Jan 19. PMID 35063702